CLINICAL TRIAL: NCT03516084
Title: A Randomized, Double-blind, Placebo-controlled, Multi-center Phase 3 Study of ZL-2306 (Niraparib) as Maintenance Therapy Following First-line Platinum-based Chemotherapy in Patients With Extensive-stage Disease Small Cell Lung Cancer (ED-SCLC) to Evaluate the Efficacy and Safety
Brief Title: A Study of Niraparib as Maintenance Therapy Following First-Line Platinum-Based Chemotherapy in Patients With Extensive Stage Small Cell Lung Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: As the treatment model of extensive-stage small cell lung cancer changed rapidly and the enrollment speed significantly lower than expected, ZaiLab decided to terminate this study
Sponsor: Zai Lab (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Zai Lab (Hong Kong), Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZL-2306-005
Record Dates: First submitted 2018-04-23; First posted 2018-05-04 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Extensive-stage Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ZL-2306(nirapairb) (Experimental)
  Interventions: Drug: ZL-2306(nirapairb)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ZL-2306(nirapairb) — The initial dose is 300mg QD or 200mg QD based on baseline weight and platelet count.
  Arms: ZL-2306(nirapairb)
Drug: Placebo — The initial dose is 300mg QD or 200mg QD based on baseline weight and platelet count.
  Arms: Placebo

SUMMARY:
Niraparib is a PARP inhibitor. The study is a 2:1 randomized, double-blind, placebo-controlled, multi-center,phase 3 study of ZL-2306 (niraparib) as maintenance therapy following first-line platinum-based chemotherapy in patients with extensive-stage disease small cell lung cancer (ED-SCLC) to evaluate the efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

Aged 18-75 years

Histologically or cytologically confirmed extensive-stage disease small cell lung cancer (ED SCLC)

Ongoing clinical benefit (partial response [PR], or complete response [CR] per RECIST version 1.1) following completion of 4 cycles of first-line platinum-based therapy (cisplatin or carboplatin, plus etoposide)

Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Subjects must have adequate bone marrow, renal and hepatic function

Exclusion Criteria:

Subjects with Central Nervous System (CNS) metastases

Subjects receiving consolidative chest radiation after last dose of first-line chemotherapy.

Subjects with pleural effusions that cannot be controlled with appropriate interventions.

All side effects attributed to prior anti-cancer therapy must have resolved to Grade 1 or baseline

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2020-02-21 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
BICR-assessed progression-free survival (PFS) | Approximately 14 months since the first subject enrolled
  The time assessed by the Blinded Independent Central Review (BICR) from randomization to progressive disease or death due to various causes, whichever occurs; progressive disease will be assessed in accordance with RECIST 1.1 criteria.
Overall survival (OS) | Approximately 48 months since first subject enrolled
  The time from randomization to death due to any cause.

SECONDARY OUTCOMES:
Investigator-assessed PFS | Approximately 14 months since the first subject enrolled
  the investigator-assessed time from randomization to progressive disease or death due to various causes, whichever occurs; progressive disease will be assessed in accordance with RECIST 1.1 criteria.

OTHER OUTCOMES:
Change in patient reported outcomes (PROs)--physical functioning domain | Approximately 48 months since first subject enrolled
  Evaluations of the quality of life of patients with small cell lung cancer include summary and analysis of absolute values and changes from baseline of various fields and single items in the patient-completed EORTC questionnaire QLQ-C30 (Version 3.0) and QLQ-LC13 Chinese version to evaluate the quality of life of lung cancer patients in the treatment group and the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Zai Lab, Study Director — Zai Lab
Locations (33):
- China (33):
  - Anhui Provincal Hospital, Hefei, Anhui
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Beijing Chest Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Cancer Hospital Chinese Academy of Medical Science, Beijing, Beijing Municipality
  - Hospital, Academy of Military Medical Sciences, Beijing, Beijing Municipality
  - Peking union medical college hospital, Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Nanfang Hospital, Guangzhou, Guangdong
  - The first affiliated hospital of Guangzhou medical school, Guangzhou, Guangdong
  - The first affiliated hospital of Guangxi Medical University, Nanning, Guangxi
  - Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - The second xiangya hospital of central south university, Changsha, Hunan
  - Nanjing General Hospital, Nanjing, Jiangsu
  - Nantong Tumor Hospital, Nantong, Jiangsu
  - The first affiliated hospital of Nanchang University, Nanchang, Jiangxi
  - The Second Affiliated hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - Jinzhou Central Hospital, Jinzhou, Liaoning
  - China shenyang chest hospital, Shenyang, Liaoning
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - Lin Yi Cancer Hospital, Linyi, Shandong
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Chest Hospital, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality
  - Tangdu Hospital, Xi’an, Shanxi
  - Xinjiang Cancer Hospital, Ürümqi, Xinjiang
  - Second Affiliated Hospital, Zhejiang University, Hangzhou, Zhejiang
  - Zhejiang cancer hospital, Hangzhou, Zhejiang
  - First Affiliated Hospital, Zhejiang University, Hanzhou, Zhejiang